CLINICAL TRIAL: NCT03918226
Title: Acute Presentation and Management of Abdominal Tuberculosis: A Ten-year Experience at a Tertiary Care Center in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Principle investigator, Services Hospital, Lahore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s16
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Tuberculosis; Abdomen
MeSH Terms: conditions — Tuberculosis | interventions — Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exploratory Laparotomy (Other): Exploratory Laparotomy of patients presenting acute abdomen and whose diagnosis later on confirmed on histopathology to be tuberculosis
  Interventions: Procedure: exploratory laparotomy

INTERVENTIONS:
Procedure: exploratory laparotomy — Patients presenting with acute abdomen were operated. Exploratory Laparotomy of patients was done. Further procedure was done according to peroperative findings. Ileostomy for perforation of gut, stricturoplasty for strictutre, biopsy for mesentric lymphadenopathy

SUMMARY:
A prospective interventional study was conducted in Services Instituton of Medical Sciences all patients who underwent emergency laparotomy from 2008-2018 due to abdominal tuberculosis. Data were analyzed using SPSS version 21

ELIGIBILITY:
Inclusion Criteria:

* Both sexes and age between years and 90 years
* Patients presenting with acute abdomen and who underwent exploratory laparotomy
* Patients who diagnosis confirmed on biopsy (caseating granulomas)

Exclusion Criteria:

* Peritoneal tuberculosis
* Other causes of acute abdomen (Typhoid perforation)
* Patients diagnosed with abdominal tuberculosis and on conservative management

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-05-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who develop complications after surgery | 9 months
  Complications of surgery like leakage of gut content, enterocutaneous fistula, intestinal obstruction
Percentage of patients who develop recurrence of abdominal tuberculosis (elevated ESR, CT scan findings of abdominal tuberculosis) | 1 year
  Recurrence of abdominal tuberclosis assessed by ESR, CT scan Abdomen, Biopsy
Mortality rate | 9 months
  death due to postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Mahmmood Ayyaz, mbbs, fcps, Study Director — Services Hospital, Lahore
Locations (1):
- Services hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided